CLINICAL TRIAL: NCT03170856
Title: The Effects of a Sub-maximal Exercise Program on Adolescents Who Sustained a Concussion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, William Meehan III, MD, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P00024907
Record Dates: First submitted 2017-05-25; First posted 2017-05-31 (Actual); Results first posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-05

CONDITIONS: Concussion, Mild; Concussion, Brain; Concussion, Severe; Exertion; Excess
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to either the exercise intervention group or the usual care group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention Group (Experimental): Thse patients will undergo a sub-maximal exercise training as treatment for concussion.
  Interventions: Other: Sub-maximal exercise
- Usual Care Group (No Intervention): These patients will not undergo a sub-maximal exercise training. They will follow the exercise instructions given to them by their physician.

INTERVENTIONS:
Other: Sub-maximal exercise — Subjects will participate in aerobic exercise 5 days a week. This includes walking, biking, jogging and running. While participating in these activities, they will be wearing their Polar Wrist Unit and Heart Rate Monitor to help subjects track their exercise intensity. They will exercise for 20 minutes 5times a week at 60% of their maximum heart rate or 80% of their symptom limited heart rate.
  Arms: Exercise Intervention Group

SUMMARY:
Patients who sustain a concussion will undergo a sub-maximal exercise protocol throughout their recovery. Cerebrovascular function, heart rate, and symptom severity, and exercise volume will be monitored throughout.

DETAILED DESCRIPTION:
There has been recent change to the management of concussion, including the addition of exercise while a patient may still be experiencing symptoms. Some patients will be given a dose-dependent exercise prescription based on their own sub-maximal output. They will aerobically exercise at this given threshold for 8 weeks, while heart rate and symptom duration is tracked. Some patients will only follow physician prescribed exercise, while undergoing the same heart rate and symptom monitoring for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Experienced a concussion within the last 2 weeks. Concussion will be diagnosed by board-certified sports medicine physicians, and defined as a direct or indirect blow to the head, face, neck, or elsewhere that manifests with the presence of symptoms and neurological impairment
* Low or moderate cardiac risk according to American College of Sports Medicine
* Post-Concussion Symptom Scale (PCSS) score greater than 9

Exclusion Criteria:

* History of neurological surgery
* Seizure disorder
* Use of medication or medical device that would alter heart rate, blood pressure or autonomic function
* Any current, serious, chronic medical or psychiatric disease that, in the Principal Investigator's judgment, may interfere with study participation or data integrity
* Unable or unwilling to provide informed consent

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2021-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Meehan, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howell DR, Taylor JA, Tan CO, Orr R, Meehan WP 3rd. The Role of Aerobic Exercise in Reducing Persistent Sport-related Concussion Symptoms. Med Sci Sports Exerc. 2019 Apr;51(4):647-652. doi: 10.1249/MSS.0000000000001829. PMID 30376513
- [Background] Howell DR, Lugade V, Taksir M, Meehan WP 3rd. Determining the utility of a smartphone-based gait evaluation for possible use in concussion management. Phys Sportsmed. 2020 Feb;48(1):75-80. doi: 10.1080/00913847.2019.1632155. Epub 2019 Jun 26. PMID 31198074
- [Background] Howell DR, Brilliant AN, Oldham JR, Berkstresser B, Wang F, Meehan WP 3rd. Exercise in the first week following concussion among collegiate athletes: Preliminary findings. J Sci Med Sport. 2020 Feb;23(2):112-117. doi: 10.1016/j.jsams.2019.08.294. Epub 2019 Sep 7. PMID 31522997
- [Background] Howell DR, Oldham J, Lanois C, Koerte I, Lin AP, Berkstresser B, Wang F, Meehan WP 3rd. Dual-Task Gait Recovery after Concussion among Female and Male Collegiate Athletes. Med Sci Sports Exerc. 2020 May;52(5):1015-1021. doi: 10.1249/MSS.0000000000002225. PMID 31985574
- [Background] Howell DR, Brilliant AN, Meehan WP 3rd. Tandem Gait Test-Retest Reliability Among Healthy Child and Adolescent Athletes. J Athl Train. 2019 Dec;54(12):1254-1259. doi: 10.4085/1062-6050-525-18. Epub 2019 Oct 28. PMID 31657636
- [Derived] Howell DR, Hunt DL, Oldham JR, Aaron SE, Meehan WP 3rd, Tan CO. Postconcussion Exercise Volume Associations With Depression, Anxiety, and Dizziness Symptoms, and Postural Stability: Preliminary Findings. J Head Trauma Rehabil. 2022 Jul-Aug 01;37(4):249-257. doi: 10.1097/HTR.0000000000000718. Epub 2021 Jul 26. PMID 34320557

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: September 1, 2018 - November 1, 2020
Period: Overall Study
Arm/Group | Exercise Intervention Group | Usual Care Group
Started | 20 | 21
Completed | 17 | 20
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: Participants who were enrolled in the study and randomized into the 2 intervention groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Intervention Group | Usual Care Group | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 14 | 25
  Between 18 and 65 years | 9 | 7 | 16
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.3 (1.9) | 16.6 (2.2) | 16.9 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 9 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 19 | 20 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 0 | 1
  White | 16 | 17 | 33
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 21 | 41

OUTCOME MEASURES:

1. Primary Outcome: Change in Vasoreactivity During Exercise at Baseline and 8-week Visits.
Description: Cerebral vasoreactivity was determined by assessing cerebrovascular conductance response to incremental hypercapnia elicited by rebreathing. Participants were fitted with a mouthpiece attached to a three-way respiratory valve unit, which, in turn, was attached to a 5-L rubber rebreathing bag. The valve allowed for an instantaneous switch from room air to the rebreathing bag, which had been prefilled with room air. EtCO2 was measured continuously via a sample line connecting the mouthpiece to an infrared CO2 analyzer.
Time Frame: Measured at initial visit and 8-weeks.
Population: Concussed participants who completed exercise testing at baseline and 8-week visits.
Measure: Mean (Standard Deviation); unit: cm s-1 mmHg-1/mmHg CO2
Groups:
- Concussed Participant Group: Participants who were enrolled in the study who were diagnosed with a sports-related concussion by a board certified sports medicine physician.
Arm/Group | Concussed Participant Group
Number analyzed (Participants) | 28
cm s-1 mmHg-1/mmHg CO2
  Baseline | 0.031 (0.013)
  8-week | 0.028 (0.010)

2. Primary Outcome: Change in Concussion Symptoms From Baseline, 4-weeks, and 8-weeks Post-injury, During an Exercise Intervention.
Description: Symptoms measured by the Post-concussion Symptom Inventory (PSCI). The PCSI ranges from 0-150 for symptom severity. The greater the number of symptoms reported, the more symptomatic the participant is. The forms focus on symptoms in the cognitive, emotional, sleep, and physical domains. There are 25 possible symptoms total. Participants answer on a scale of 0-6 for symptom severity (0- not a problem, 3- moderate problem, 6- severe problem).
Time Frame: The PSCI symptom severity be a repeated measured at the time of injury, 4 weeks post-injury and 8 weeks post-injury, to look for a change in symptom score over the duration of the study.
Population: Those who reported sufficient exercise volume information during the duration of the study.
Measure: Median (Inter-Quartile Range); unit: score on the PSCI scale
Groups:
- Exercise Intervention Group: These patients will undergo a sub-maximal exercise training as treatment for concussion.
  Sub-maximal exercise: Subjects will participate in aerobic exercise 5 days a week. This includes walking, biking, jogging and running. While participating in these activities, they will be wearing their Polar Wrist Unit and Heart Rate Monitor to help subjects track their exercise intensity. They will exercise for 20 minutes 5times a week at 60% of their maximum heart rate or 80% of their symptom limited heart rate.
Arm/Group | Exercise Intervention Group | Usual Care Group
Number analyzed (Participants) | 17 | 19
score on the PSCI scale
  Initial | 15 [10 to 42] | 20 [11 to 35.5]
  4weeks post injury | 4 [0 to 28] | 5.5 [0.5 to 21.5]
  8weeks post injury | 6.5 [0 to 27.5] | 0 [0 to 4]

3. Secondary Outcome: End-tidal CO2
Description: Will be monitored using infrared analyzer during sub-maximal exercise testing at baseline and 8-week post injury visits.
Time Frame: Measured at initial visit and 8-week post injury visit.
Population: Participants enrolled in the study who completed exercise testing sessions at baseline and 8-week post injury.
Measure: Mean (Standard Deviation); unit: mmHG
Arm/Group | Concussed Participant Group
Number analyzed (Participants) | 25
mmHG
  Baseline | 33.4 (3.0)
  8-week | 33.2 (2.6)

4. Secondary Outcome: Heart Rate
Description: Monitored via standard 3 lead ECG during sub-maximal exercise testing at initial and 8-week visits.
Time Frame: Measured at initial visit and 8 weeks to look for a change as a person becomes asymptomatic.
Population: Participants who completed exercise testing at baseline, 4-week, and 8-week follow-up visits.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Exercise Intervention Group | Usual Care Group
Number analyzed (Participants) | 17 | 19
beats per minute (bpm)
  Baseline Baseline | 162.5 (19) | 164.5 (14.9)
  4-Week | 171.1 (9.6) | 170 (9.8)
  8-Week | 170.2 (8.1) | 167.4 (12.3)

5. Secondary Outcome: Volume of Self-reported Exercise Per Week
Description: Volume exercise was monitored by self-reported exercise diary. All participants were asked to track their exercise and complete weekly exercise logs for the 8-week study duration. The participants randomized into the Exercise Intervention Group were prescribed a specific heart rate to exercise 5x/week for 8-weeks. Heart rate was determined by their performance from the corresponding exercise testing visit. Participants enrolled in the Usual Care Group were not prescribed any specific exercise. These participants were instructed to follow their Doctors requests. Values are presented as average minutes of exercise throughout the 8-week study period.
Time Frame: Average volume of exercise (min) that was self-reported by participants over the 8-week study period.
Population: Those who reported sufficient exercise volume information during the duration of the study.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Exercise Intervention Group | Usual Care Group
Number analyzed (Participants) | 17 | 20
minutes | 115 [54 to 225] | 88 [28 to 230]

6. Secondary Outcome: Rate of Perceived Exhaustion at Baseline, 4-week, and 8-week Visits.
Description: Using the Borg Scale. The Borg scale is a way of measuring physical intensity level. The scale ranges from 6- no exertion at all, to 20- maximal exertion. The higher the RPE reported, the harder the participant perceives themselves to be physically working.
Time Frame: Measured at initial visit, 4 weeks and 8 weeks to look for a change in perceived exhaustion as a person becomes asymptomatic
Population: Those who reported RPE during initial, 4-week, and 8-week exercise tests.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise Intervention Group | Usual Care Group
Number analyzed (Participants) | 17 | 19
units on a scale
  baseline | 15.8 (2.3) | 15.4 (1.7)
  4-Week | 16.7 (1.8) | 15.5 (1.9)
  8-Week | 16.7 (1.9) | 15.1 (2.1)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout each participant's enrollment in the study. This included at their initial visit, 4-weeks post injury, and 8-weeks post injury.
Arm/Group | Exercise Intervention Group | Usual Care Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT03170856/Prot_SAP_000.pdf